CLINICAL TRIAL: NCT00136981
Title: Phase 3 Multi-Center, Double-Blind, Randomized, Parallel Group, Carotid B-Mode Ultrasound Evaluation of the Anti-Atherosclerotic Efficacy, Safety and Tolerability of Fixed Combination CP-529,414/Atorvastatin, Administered Orally, Once Daily (QD) for 24 Months, Compared With Maximally Tolerated Atorvastatin Therapy Alone, in Subjects With Heterozygous Familial Hypercholesterolemia.
Brief Title: Carotid B-Mode Ultrasound Study to Compare Anti-Atherosclerotic Effect of Torcetrpib/Atorvastatin to Atorvastatin Alone.
Acronym: RADIANCE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5091003
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Hypercholesterolemia, Familial; Hyperlipidemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hyperlipidemias | interventions — torcetrapib; Atorvastatin

INTERVENTIONS:
Drug: torcetrapib/atorvastatin
Drug: atorvastatin

SUMMARY:
The Torcetrapib project was terminated on December 2, 2006 due to safety findings.

To look at ultrasound images taken in the carotid arteries and to look at various lipids in the blood of people with heterozygous familial hypercholesterolemia

DETAILED DESCRIPTION:
For additional information please call: 1-800-718-1021

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Heterozygous Familial Hypercholesterolemia
* At least 18 years of age

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant.
* Subjects with a clinically indicated need for statin (HMG-CoA reductase inhibitor) therapy other than atorvastatin or other concomitant therapy with known lipid altering effects on LDL-C and HDL-C including fibrates and nicotinic acid (high doses)
* Subjects taking any drugs known to be associated with an increased risk of myositis in combination with HMG-CoA reductase inhibitors
* Subjects with any other medical condition or laboratory abnormality which could affect subject safety, preclude evaluationof response, or render unlikely that the subject would complete the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2003-12; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change in intima media thickness as measures by carotid ultrasound

SECONDARY OUTCOMES:
Changes in levels of lipids and other biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (34):
- United States (7):
  - Pfizer Investigational Site, Hartford, Connecticut
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Seattle, Washington
- Canada (5):
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
- Pfizer Investigational Site, Prague, Czechia
- Finland (2):
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, OYS
- France (2):
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Toul
- Italy (2):
  - Pfizer Investigational Site, Brescia
  - Pfizer Investigational Site, Pavia
- Netherlands (12):
  - Pfizer Investigational Site, Alkmaar
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Delft
  - Pfizer Investigational Site, Goes
  - Pfizer Investigational Site, Groningen
  - Pfizer Investigational Site, Hoorn
  - Pfizer Investigational Site, Leiden
  - Pfizer Investigational Site, Nijmegen
  - Pfizer Investigational Site, Rotterdam
  - Pfizer Investigational Site, Sliedrecht
  - Pfizer Investigational Site, Utrecht
  - Pfizer Investigational Site, Waalwijk
- South Africa (3):
  - Pfizer Investigational Site, Parow, Cape Town
  - Pfizer Investigational Site, Parktown, Johannesburg
  - Pfizer Investigational Site, Cape Town

REFERENCES:
- [Derived] Tajik P, Meijer R, Duivenvoorden R, Peters SA, Kastelein JJ, Visseren FJ, Crouse JR 3rd, Palmer MK, Raichlen JS, Grobbee DE, Bots ML. Asymmetrical distribution of atherosclerosis in the carotid artery: identical patterns across age, race, and gender. Eur J Prev Cardiol. 2012 Aug;19(4):687-97. doi: 10.1177/1741826711410821. Epub 2011 May 25. PMID 21613319
- [Derived] Dogan S, Duivenvoorden R, Grobbee DE, Kastelein JJ, Shear CL, Evans GW, Visseren FL, Bots ML; Radiance 1 and Radiance 2 Study Groups. Ultrasound protocols to measure carotid intima-media thickness in trials; comparison of reproducibility, rate of progression, and effect of intervention in subjects with familial hypercholesterolemia and subjects with mixed dyslipidemia. Ann Med. 2010 Sep;42(6):447-64. doi: 10.3109/07853890.2010.499132. PMID 20645885
- [Derived] Dogan S, Duivenvoorden R, Grobbee DE, Kastelein JJ, Shear CL, Evans GW, Visseren FL, Bots ML; Radiance 1 and 2 Study Groups. Completeness of carotid intima media thickness measurements depends on body composition: the RADIANCE 1 and 2 trials. J Atheroscler Thromb. 2010 May;17(5):526-35. doi: 10.5551/jat.3269. Epub 2010 Mar 13. PMID 20228610
- [Derived] Vergeer M, Bots ML, van Leuven SI, Basart DC, Sijbrands EJ, Evans GW, Grobbee DE, Visseren FL, Stalenhoef AF, Stroes ES, Kastelein JJ. Cholesteryl ester transfer protein inhibitor torcetrapib and off-target toxicity: a pooled analysis of the rating atherosclerotic disease change by imaging with a new CETP inhibitor (RADIANCE) trials. Circulation. 2008 Dec 9;118(24):2515-22. doi: 10.1161/CIRCULATIONAHA.108.772665. Epub 2008 Nov 24. PMID 19029469
- [Derived] Kastelein JJ, van Leuven SI, Evans GW, Riley WA, Revkin JH, Shear CL, Bots ML; RADIANCE 1 and 2 Study Investigators. Designs of RADIANCE 1 and 2: carotid ultrasound studies comparing the effects of torcetrapib/atorvastatin with atorvastatin alone on atherosclerosis. Curr Med Res Opin. 2007 Apr;23(4):885-94. doi: 10.1185/030079907x182121. PMID 17407645
- [Derived] Kastelein JJ, van Leuven SI, Burgess L, Evans GW, Kuivenhoven JA, Barter PJ, Revkin JH, Grobbee DE, Riley WA, Shear CL, Duggan WT, Bots ML; RADIANCE 1 Investigators. Effect of torcetrapib on carotid atherosclerosis in familial hypercholesterolemia. N Engl J Med. 2007 Apr 19;356(16):1620-30. doi: 10.1056/NEJMoa071359. Epub 2007 Mar 26. PMID 17387131
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5091003&StudyName=Carotid+B%2DMode+Ultrasound+Study+to+Compare+Anti%2DAtherosclerotic+Effect+of+Torcetrpib%2FAtorvastatin+to+Atorvastatin+Alone%2E